CLINICAL TRIAL: NCT01646502
Title: Treatment of Chronic Wound Staphylococcus Aureus Biofilms With Staphylococcus Epidermidis Esp Protein to Promote Healing
Brief Title: Treatment of Chronic Wound Biofilms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was discontinued. Ran into difficulties with purification at the protein production stage
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H12-00862
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Wound; Venous Insufficiency; Biofilms
Keywords: chronic wound; treatment; biofilms; venous insufficiency; Esp
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esp-supplemented standard wound care (Experimental): 500 pmol Esp protein will be added to the standard wound care protocol.
  Interventions: Biological: Esp protein
- Standard wound care (Active Comparator): The standard treatment protocol established at the Vancouver Wound Healing Clinic is based on the "Best Clinical Practice Guidelines for Venous Leg Ulcers" from the Canadian Association of Wound Care.
  Interventions: Other: Standard wound care

INTERVENTIONS:
Biological: Esp protein
  Arms: Esp-supplemented standard wound care
Other: Standard wound care
  Arms: Standard wound care

SUMMARY:
Chronic wounds cause significant morbidity and cost our healthcare system millions of dollars each year.Their healing is slowed by biofilms, communities of bacteria surrounded by a protective layer that stops the immune system and antibiotics from getting close enough to kill them. The investigators will develop a new strategy to destroy biofilms using a protein made from bacteria that live on our skin.The Staphylococcus epidermidis Esp protein will be used to destroy Staphylococcus aureus biofilms, the most common bacterium in chronic wounds. The investigators hypothesize that the use of the Esp protein will breakdown S. aureus biofilms, decrease bacterial colonization of chronic wounds and improve healing times.

DETAILED DESCRIPTION:
Chronic wounds lead to significant patient morbidity and mortality, and its treatment is associated with a global economic burden of $13-$15 billion annually. In Canada, the average cost of three months of community care for a chronic wound is $ 27,600.00. One of the major complications associated with chronic wounds is colonization with a Staphylococcus aureus (S. aureus) biofilm. These bacterial biofilms delay re-epithelialization and prevent wound healing. Standard treatment of chronic wound biofilms includes aggressive debridement as well as the addition of anti-biofilm agents such as antimicrobials. Since antimicrobial resistance is becoming a serious problem, finding alternatives is essential.

Staphylococcus epidermidis (S. epidermidis) JK16 cells, their culture supernatants and a serine protease (Esp) in the culture supernatants have been shown to inhibit the formation of and destroy preexisting S. aureus biofilms. The investigators hypothesize that the use of S. epidermidis JK16, culture supernatants or purified Esp protein in the standard wound care protocol will breakdown S. aureus biofilms, decrease bacterial colonization of chronic wounds and improve healing times. The investigators will employ a two-way cross over study where participants will receive standard wound care or S. epidermidis JK16 Esp supplemented treatment for the first 6 weeks followed by cross over for a further 6 weeks. These patients will be recruited from the Wound Healing Clinic at Vancouver General Hospital. Standard wound care will be provided in accordance with established protocols based on "Best Clinical Practice Guidelines for Venous Leg Ulcers" from the Canadian Association of Wound Care. For the S. epidermidis JK16 Esp supplemented treatment arm, the investigators will produce purified Esp and impregnate wound dressings with this protein. After 6 weeks, participants will be crossed over to the corresponding treatment arm.

Our primary outcome measure will be healing rate as calculated for each 6 week standard or experimental treatment periods. The investigators will employ standardized photography and wound image analysis software to calculate the healing rate. Other outcome measures will include visual detection and qualitative assessment of biofilms as determined by trained nurses and/or physicians. Finally, bacterial type and quantity will be determined by wound biopsy. Outcome measures for standard treatment arms will be compared with results from S. epidermidis JK16 Esp supplemented treatment arms. Objectives of this pilot study include:

1. To assess the feasibility of conducting a more definitive trial to examine the efficacy of S. epidermidis Esp protein from strain JK16 in healing chronic wounds
2. To perform a pilot study using a cross-over design with the purified S. epidermidis Esp protein from strain JK16 in comparison to standard therapy
3. To demonstrate that the intervention is acceptable to participants
4. To demonstrate the safety of the intervention
5. To explore the biologic activity of S. epidermidis Esp protein from strain JK16 on wound biofilms and healing times

ELIGIBILITY:
Inclusion Criteria:

1. Have a leg ulcer with the ankle brachial pressure index (ABPI) equal or greater than 0.6;
2. Have a wound that is 15 cm or less in diameter;
3. Are 19 years or older;
4. Have no known contraindication to the treatment products

Exclusion Criteria:

1. Have a leg ulcer caused by pressure, diabetes, ischemia, inflammatory disorder, hematologic disorder or malignancy
2. Have applied an antiseptic to the wound in the one week prior to recruitment
3. Have received systemic or topical antibiotic therapy within 48 hours prior to recruitment
4. Are being treated with systemic steroids (prednisone)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
rate of wound healing | 6 weeks
  The rate of wound healing (% change in wound surface area) over each 6-week treatment period.

SECONDARY OUTCOMES:
A qualitative assessment of the healing process. | 1 week
  A physician or nurse will record a visual assessment of the chronic wound in order to obtain a qualitative wound score.

OTHER OUTCOMES:
Bacterial type and quantity. | 6 weeks
  This will be determined by wound biopsy performed at baseline and at weeks 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kunimoto, MD, Principal Investigator — University of British Columbia
Locations (1):
- Wound Healing Clinic,Vancouver General Hospital - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada